CLINICAL TRIAL: NCT04384120
Title: Use of Blood Flow Restriction (BFR) Therapy in Patients With Rotator Cuff Tears Treated Nonoperatively or Operatively: a Randomized Controlled Trial
Brief Title: BFR Therapy in Patients With Rotator Cuff Tears
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Patient Follow-up
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Vasilios Moutzouros, Orthopedic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13130
Record Dates: First submitted 2020-05-01; First posted 2020-05-12 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Blood Flow Restriction
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Rotator Cuff Rehabilitation Using BFR (Experimental): Patients with rotator cuff tears who plan for either nonoperative treatment with physical therapy or operative treatment with arthroscopic rotator cuff repair (RCR) surgery will be randomized to undergo rehabilitation using blood flow restriction cuffs.
  1. Patients who elect for nonoperative treatment of their rotator cuff tear will undergo traditional therapy using blood flow restriction cuffs.
  2. Patients who elect for RCR will undergo preoperative and postoperative traditional therapy using blood flow restriction cuffs.
  Interventions: Device: Blood Flow Restriction Therapy
- Rotator Cuff Rehabilitation Without BFR (Active Comparator): Patients with rotator cuff tears who plan for either nonoperative treatment with physical therapy or operative treatment with arthroscopic rotator cuff repair (RCR) surgery will be randomized to undergo rehabilitation without using blood flow restriction cuffs.
  1. Patients who elect for nonoperative treatment of their rotator cuff tear will undergo traditional therapy without using blood flow restriction cuffs.
  2. Patients who elect for RCR will undergo preoperative and postoperative traditional therapy without using blood flow restriction cuffs.
  Interventions: Procedure: Traditional Therapy

INTERVENTIONS:
Device: Blood Flow Restriction Therapy — Blood flow restriction cuffs which are FDA approved will be provided to patients randomized into the BFR group. Patients will be provided video instruction and training on how to conduct the traditional therapy exercises with the use of BFR.
  Arms: Rotator Cuff Rehabilitation Using BFR
Procedure: Traditional Therapy — Patients will be provided video instruction and training on how to conduct the traditional therapy exercises.
  Arms: Rotator Cuff Rehabilitation Without BFR

SUMMARY:
The purpose of this study is to examine the effect of utilizing blood flow restriction (BFR) therapy in patients treated both non operatively and operatively for rotator cuff tears (RCT). BFR has been proposed to work by restricting arterial inflow leading to an oxygen depleted environment and the ability to induce muscle adaption at lower maximum repetition via reactive hyperemia. Muscle atrophy occurs following rotator cuff tear. Thus, physical therapy is used to regain strength with the ultimate goal of returning to activity.

The goal of this investigation is to determine if using BFR during therapy for non-operatively managed and operatively managed rotator cuff tears would lead to increased and expedited strength gains. Additionally the investigators would like to determine if BFR is beneficial in preventing muscle atrophy and fatty infiltration often seen in the setting of rotator cuff tear, as it is known that cuff tears can subject the muscles to degenerative changes and these patients are at risk for poorer clinical outcomes. The investigators will also look at patient reported outcomes metrics and pain scores to determine if BFR has a significant impact on the patient experience surrounding rotator cuff tear after both nonoperative treatment with therapy and operative treatment with surgical repair and peri-operative rehabilitation.

The investigators hypothesize that the BFR group will have significantly greater strength gains at all time points. Previous studies have shown that BFR has potential in increasing muscle torque generation and cross sectional area in the first six months following anterior cruciate ligament (ACL) reconstruction. While there have not been as many studies investigating the use of BFR following upper extremity surgery, previous research has demonstrate that BFR can be useful both proximal and distal to the targeted muscle groups in the upper extremity. In addition to the paucity of research on post-operative BFR following rotator cuff repair (RCR), there is no evidence on pre-operative use as well. The investigators believe that the use of BFR in the perioperative period surrounding rotator cuff tear and repair has the potential to significantly decrease muscle atrophy and lead to faster, more substantial strength gains and less muscle atrophy and fatty infiltration.

DETAILED DESCRIPTION:
Patients who are seen in clinic for rotator cuff pathology will undergo treatment for their rotator cuff based on a shared-decision making process with the orthopedic surgeon, irrespective of this study. Once a treatment plan is in place, the patient will be introduced to this study and presented with the opportunity to participate. If the patient agrees, a formal consent process will take place in clinic and the patient will undergo initial, baseline testing of strength, range of motion, pain scores, and patient reported outcome scores.

Therefore patients will be either in the nonoperative arm or the operative arm of this study. Within each arm, patients will be randomized via computer to be placed in either the blood flow restriction (BFR) cohort or the traditional (non-BFR cohort). Patients will prospectively undergo rotator cuff rehabilitation using BFR or conventional therapy by physical therapists with extensive experience in rotator cuff rehabilitation who will undergo training on use of BFR.

The nonoperative group will be given identical rehabilitation protocols, with the only difference being the use of a BFR cuff during rehabilitation for the BFR cohort. Similarly, the operative group will be given identical rehabilitation protocols, with the only difference being the use of a BFR cuff during rehabilitation for the BFR cohort.

Patients undergoing operative rotator cuff repair (RCR) will undergo preoperative rehabilitation prior to surgery for two weeks. Due to limitations of health insurance coverage of physical therapy sessions, the two weeks of preoperative "prehab" will consist of a structured home exercise program that is taught to the patient by a physical therapist during one session and recorded on a physical therapy (PT) diary by the patient during the two weeks leading up to surgery. Patients will be provided video instruction and training on how to conduct the exercises and this will also be done with and without the use of BFR depending on group allocation (via randomization). Additionally, warning signs for BFR cuff intolerance such as increased pain, swelling, numbness/tingling of the arm will be communicated to the patient. Following surgery patients will immediately be started in a formal physical therapy regimen as an outpatient. Therapy will consist of a structured program progressing from range of motion, to strength training and then functional tests. Patients will remain in their allocated BFR or non-BFR group.

Protocol as follows, both groups will use the same protocol with the only difference being use of BFR:

For surgical patients:

• Preop: Patients will undergo a home program consisting of isometric exercises including shoulder extension, abduction, external rotation and internal rotation pushing against a wall.

For both surgical and non-surgical patients:

* Post-op weeks 0-8: Passive shoulder range of motion (ROM) only

  * Sling immobilization with active elbow, wrist and hand ROM
  * Passive ROM only of shoulder including pendulums, supine elevation in scapular plane, external rotation with arm at side.
* 8-12 weeks being more active range of motion

  * Discontinue sling
  * Being active exercises including prone row, standing internal/external rotation with bands, wall slides into shoulder flexion
* Weeks 12-20: Strength and function o Sidelying shoulder external rotation, increase resistance band exercises

Throughout this protocol patients will have a pre-operative visit, an early 2 week post operative visit to check range of motion and wound healing, a six week visit to monitor range of motion and potentially clear for active ROM and sling discontinuation, and a three month visit prior to clearance to being return to more aggressive activity. Strength and range of motion will be recorded at each of these visits in order to assess the primary endpoint.

Outcomes:

* Primary Outcome:

  o Strength to be measured via dynamometer at each clinic visit
* Secondary Outcomes:

  * Range of motion via goniometer
  * Pain via visual analogue scale (VAS) pain scale at each visit
  * Patient reported outcomes scores at each visit
  * Fatty infiltration and muscle atrophy measured via ultrasound and compared to pre-operative imaging

Plan to recruit patients starting in June 2020. Will enroll patients and collect data from June-2020 to May 2021. Manuscript writing and submission to occur in June 2021.

* Data analysis: The primary endpoint of this study was a maximum repetition total work deficit of 15% between the BFR and control group as measured by dynamometer. This was based on previous data showing that a strength deficit of 15% represents a clinically significant difference that is not likely attributable to limb dominance. Work deficit was calculated in each group by comparing the operative leg with the nonoperative leg to obtain a deficit percent. A power analysis was performed before the study to assess the number of patients needed to detect a 15% total work deficit between the BFR and control groups. With a power of 80% (beta level ¼ 0.80, alpha level ¼ 0.05), a sample size of 34 (17 patients per group) was obtained. Data will be provided to and analyzed by trained statisticians to determine differences in primary and secondary outcomes.
* All continuous data will be analyzed using independent 2-group t tests and reported as means ± standard deviations. Categorical data will be compared between the 2 groups using chi-square tests and reported as counts and percentages. A preliminary test to confirm the quality of variances will be conducted prior to utilizing the t test to confirm the appropriate statistical analysis. Nonparametric equivalents Wilcoxon rank-sum and Fisher exact tests will be used as needed for nonnormal distributions and low variable numbers, respectively. A multivariable regression analysis was performed to assess for potential confounding demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-80 who suffered a rotator cuff tear
* Patients undergoing arthroscopic rotator cuff repair
* Patients undergoing nonoperative treatment with physical therapy

Exclusion Criteria:

* Subjects will be excluded if they are undergoing revision rotator cuff repair, history of DVT, neurovascular injury, unable to tolerate BFR treatment, unable to complete physical therapy, peripheral vascular disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lafi S Khalil, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
per request

REFERENCES:
- [Background] Clark BC, Manini TM, Hoffman RL, Williams PS, Guiler MK, Knutson MJ, McGlynn ML, Kushnick MR. Relative safety of 4 weeks of blood flow-restricted resistance exercise in young, healthy adults. Scand J Med Sci Sports. 2011 Oct;21(5):653-62. doi: 10.1111/j.1600-0838.2010.01100.x. Epub 2010 Mar 11. PMID 21917016
- [Background] Dankel SJ, Jessee MB, Abe T, Loenneke JP. The Effects of Blood Flow Restriction on Upper-Body Musculature Located Distal and Proximal to Applied Pressure. Sports Med. 2016 Jan;46(1):23-33. doi: 10.1007/s40279-015-0407-7. PMID 26446893
- [Background] Hamano N, Yamamoto A, Shitara H, Ichinose T, Shimoyama D, Sasaki T, Kobayashi T, Kakuta Y, Osawa T, Takagishi K. Does successful rotator cuff repair improve muscle atrophy and fatty infiltration of the rotator cuff? A retrospective magnetic resonance imaging study performed shortly after surgery as a reference. J Shoulder Elbow Surg. 2017 Jun;26(6):967-974. doi: 10.1016/j.jse.2016.10.016. Epub 2017 Feb 15. PMID 28214172
- [Background] Kuzel BR, Grindel S, Papandrea R, Ziegler D. Fatty infiltration and rotator cuff atrophy. J Am Acad Orthop Surg. 2013 Oct;21(10):613-23. doi: 10.5435/JAAOS-21-10-613. PMID 24084435
- [Background] Madarame H, Sasaki K, Ishii N. Endocrine responses to upper- and lower-limb resistance exercises with blood flow restriction. Acta Physiol Hung. 2010 Jun;97(2):192-200. doi: 10.1556/APhysiol.97.2010.2.5. PMID 20511128
- [Background] Melis B, DeFranco MJ, Chuinard C, Walch G. Natural history of fatty infiltration and atrophy of the supraspinatus muscle in rotator cuff tears. Clin Orthop Relat Res. 2010 Jun;468(6):1498-505. doi: 10.1007/s11999-009-1207-x. PMID 20094853
- [Background] Noordin S, McEwen JA, Kragh JF Jr, Eisen A, Masri BA. Surgical tourniquets in orthopaedics. J Bone Joint Surg Am. 2009 Dec;91(12):2958-67. doi: 10.2106/JBJS.I.00634. PMID 19952261
- [Background] Ohta H, Kurosawa H, Ikeda H, Iwase Y, Satou N, Nakamura S. Low-load resistance muscular training with moderate restriction of blood flow after anterior cruciate ligament reconstruction. Acta Orthop Scand. 2003 Feb;74(1):62-8. doi: 10.1080/00016470310013680. PMID 12635796
- [Background] Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc. 2000 Dec;32(12):2035-9. doi: 10.1097/00005768-200012000-00011. PMID 11128848
- [Background] Wernbom M, Augustsson J, Raastad T. Ischemic strength training: a low-load alternative to heavy resistance exercise? Scand J Med Sci Sports. 2008 Aug;18(4):401-16. doi: 10.1111/j.1600-0838.2008.00788.x. Epub 2008 May 3. PMID 18466185

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotator Cuff Rehabilitation Using BFR: Patients with rotator cuff tears who plan for either nonoperative treatment with physical therapy or operative treatment with arthroscopic rotator cuff repair (RCR) surgery will be randomized to undergo rehabilitation using blood flow restriction cuffs.
  1. Patients who elect for nonoperative treatment of their rotator cuff tear will undergo traditional therapy using blood flow restriction cuffs.
  2. Patients who elect for RCR will undergo preoperative and postoperative traditional therapy using blood flow restriction cuffs.
  Blood Flow Restriction Therapy: Blood flow restriction cuffs which are FDA approved will be provided to patients randomized into the BFR group. Patients will be provided video instruction and training on how to conduct the traditional therapy exercises with the use of BFR.
- Rotator Cuff Rehabilitation Without BFR: Patients with rotator cuff tears who plan for either nonoperative treatment with physical therapy or operative treatment with arthroscopic rotator cuff repair (RCR) surgery will be randomized to undergo rehabilitation without using blood flow restriction cuffs.
  1. Patients who elect for nonoperative treatment of their rotator cuff tear will undergo traditional therapy without using blood flow restriction cuffs.
  2. Patients who elect for RCR will undergo preoperative and postoperative traditional therapy without using blood flow restriction cuffs.
  Traditional Therapy: Patients will be provided video instruction and training on how to conduct the traditional therapy exercises.
Period: Overall Study
Arm/Group | Rotator Cuff Rehabilitation Using BFR | Rotator Cuff Rehabilitation Without BFR
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotator Cuff Rehabilitation Using BFR | Rotator Cuff Rehabilitation Without BFR | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10) | 55.9 (6) | 58.2 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Strength [Mean (Standard Deviation); unit: Pounds] — Measured by Dynamometer
  Pounds | 7.34 (4.14) | 7.24 (4.14) | 7.3 (3.23)

OUTCOME MEASURES:

1. Primary Outcome: Strength
Description: Strength will be quantified through dynamometers
Time Frame: through study completion, an average of 12 months post-operative follow-up
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Rotator Cuff Rehabilitation Using BFR | Rotator Cuff Rehabilitation Without BFR
Number analyzed (Participants) | 15 | 15
Pounds | 7.39 (3.93) | 6.05 (3.1)

2. Secondary Outcome: Range of Motion
Description: Range of motion of the shoulder will be assessed using a goniometer
Time Frame: through study completion, an average of 12 months post-operative follow-up
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rotator Cuff Rehabilitation Using BFR | Rotator Cuff Rehabilitation Without BFR
Number analyzed (Participants) | 15 | 15
degrees | 82.4 (24.7) | 65.1 (18.8)

3. Secondary Outcome: Pain Score
Description: Pain will be assessed using a visual analogue scale (VAS), a pain scale from 0-10 where higher numbers indicate worse pain
Time Frame: through study completion, an average of 12 months post-operative follow-up
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Rotator Cuff Rehabilitation Using BFR | Rotator Cuff Rehabilitation Without BFR
Number analyzed (Participants) | 15 | 15
points | 30.3 (4.7) | 26.3 (6.3)

4. Secondary Outcome: Patient Reported Outcomes Measurement Information System
Description: Patient reported outcome measurement information system (PROMIS) scores will be collected through a series of questionnaires from the PROMIS domain of physical function, upper extremity, and depression. These scores are standardized T-scores with the mean set at 50 and the standard deviation set at 10.
  PROMIS scores for Physical function, the higher the score the better. PROMIS score for depression, the lower the score the better. PROMIS score for Upper extremity, the higher the score the better.
Time Frame: through study completion, an average of 12 months post-operative follow-up
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Rotator Cuff Rehabilitation Using BFR | Rotator Cuff Rehabilitation Without BFR
Number analyzed (Participants) | 15 | 15
points
  PROMIS-UE | 30.3 (4.7) | 26.3 (6.3)
  PROMIS-PI | 63 (8.8) | 63 (6.7)
  PROMIS-D | 47 (9.8) | 47 (9.4)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Rotator Cuff Rehabilitation Using BFR | Rotator Cuff Rehabilitation Without BFR
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04384120/Prot_SAP_001.pdf